CLINICAL TRIAL: NCT05507554
Title: Effectiveness of Different Postoperative Analgesics Use in the Management of Acute Pain After Ureteroscopy.
Brief Title: Different Postoperative Analgesics Use After Ureteroscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pakistan Kidney and Liver Institute and Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PKLI Nadeem Iqbal
Record Dates: First submitted 2022-08-17; First posted 2022-08-19 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Post Operative Pain; Ureteroscopy; Ureter Stone
Keywords: Pain; Analgesics; Non-Steroidal; Opioid; Urolithiasis; Ureteroscopy
MeSH Terms: conditions — Pain, Postoperative; Ureterolithiasis; Pain; Urolithiasis | interventions — Analgesics, Opioid; Analgesics, Non-Narcotic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Opioid Group (Active Comparator): This group comprises of patients with ureter stones stones who undergo ureteroscopy procedure. They will be randomized to intravenous injection Tramadol 50 mg. They will also be discharged on Tramadol oral capsule 50 mg for postoperative pain after the ureteroscopy procedure with stent placement
  Interventions: Drug: Opioid
- Paracetamol (Acetaminophen) Group (Active Comparator): This group comprises of patients with ureter stones stones who undergo ureteroscopy procedure. They will be randomized to intravenous injection Paracetamol 1 Gram. They will also be discharged on oral Tablet Paracetamol 1 Gram for postoperative pain after the ureteroscopy procedure with stent placement
  Interventions: Drug: Non-Opioid Analgesic
- Diclofenac Sodium Group (Active Comparator): This group comprises of patients with ureter stones stones who undergo ureteroscopy procedure. They will be randomized to intra muscular injection Diclofenac Sodium 50 mg. They will also be discharged on oral Tablet Diclofenac Sodium 50 mg for postoperative pain after the ureteroscopy procedure with stent placement.
  Interventions: Drug: Non-Opioid

INTERVENTIONS:
Drug: Opioid — Drug: intravenous injection Tramadol 50 mg and then oral capsule Tramadol 50 mg, once patient starts taking orally.
  Designated coated 14 days supply of pain medication (oral capsule Tramadol 50 mg) will be given to the patients on discharge. For Pain control oral capsule Tramadol 50 mg is administered 2 times per day until the stent will be removed in clinic 2 weeks later.
  Arms: Opioid Group
Drug: Non-Opioid Analgesic — Drug: intravenous injection Paracetamol 1 Gram and then oral Tablet Paracetamol 1 Gram, once patient starts taking orally.
  Designated coated 14 days supply of pain medication (oral Tablet Paracetamol 1 Gram) will be given to the patients on discharge. For Pain control oral Paracetamol 1 Gram is administered 3 times per day until the stent will be removed in clinic 2 weeks later.
  Arms: Paracetamol (Acetaminophen) Group
Drug: Non-Opioid — Drug: intra muscular injection Diclofenac Sodium 50 mg and then oral Tablet Diclofenac Sodium 50 mg, once patient starts taking orally.
  Designated coated 14 days supply of pain medication (oral Tablet Diclofenac Sodium 50 mg) will be given to the patients on discharge. For Pain control oral Diclofenac Sodium 50 mg is administered 2 times per day until the stent will be removed in clinic 2 weeks later.
  Arms: Diclofenac Sodium Group

SUMMARY:
In this study, we will see the feasibility of a non-opioid pain killers in management of acute post-operative period as well as on discharge from the hospital compared to opioid medications for postoperative pain following URS and stent placement.

The objective of this study will be to compare the pain control effects of no opioid and opioid pain killers during the post-operative period. This study will be a Randomized Clinical trial. Data will be collected from department of Urology, PKLI, Lahore. All patients included in this study will undergo ureteroscopic laser lithotripsy of ureter stones. One group will receive tramadol (opioid) while other two groups will receive Paracetamol and diclofenac sodium (NSAIDs) respectively. All subjects will receive one of the three pain killers after ureteroscopy procedure for ureter stones in a randomized fashion. Postoperative pain intensity will be measured by the investigator and the nurse in the first hour after the surgery in the recovery room and then in urology ward at 1,6, 12, 24, 48, & 72 hours using the Numeric Pain Intensity Scale (NPIS).A mean pain score of less than 2 for each category of surgical procedures or analgesics group will be defined as satisfactory pain control. The data will be analyzed using SPSS v 24.

DETAILED DESCRIPTION:
Achieving adequate postoperative pain relief should be a definitive goal of patient care in any surgery because pain is one of the most common postoperative symptoms as reported from previous studies. Efforts have begun to implement non opioid protocols for outpatient urologic surgery. Recently it was found that Ureteroscopy (URS) with stent placement is possible without using postoperatve opioids for pain control and stent-related symptoms. To date, attention has focused on the problems of opioid abuse, diversion, and overdose. These issues pertain primarily to those who are already suffering from substance use disorders. More recently, the possibility that legitimate use of prescription opioids has led to incident substance use disorders (iatrogenic addiction) is beginning to gather attention.

When iatrogenic addiction has been considered, it is almost exclusively in the context of chronic pain. Not surprisingly, emergency providers commonly believe that short courses of opioid therapy for acute pain are safe and that their role in the current opioid crisis is limited to attenuating diversion. However, several recent studies have demonstrated that short course opioid therapy for acute pain is associated with future recurrent use of opioids, raising the possibility that short course opioid therapy may be a potential trigger for the onset of opioid related substance use disorders. If so, there are considerable health implications as more than 1 in every 6 patients discharged from an ED are given a prescription for an opioid pain reliever.

In this study, we will see the feasibility of a non-opioid discharge protocol compared to standard opioid medications for postoperative pain following URS and stent placement. We will also evaluate the effect of these analgesic in acute pain management in post op stay in hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Ureteroscopy procedure performed for ureteric stones between age 18 -60 years.
2. Patients with normal Renal and Liver function tests function tests.
3. Patients having no growth on urine culture will be included in this study.
4. Patients with no previous history of ureteroscopy procedure in past.

Exclusion Criteria:

1. Patients having history of allergic reaction to any type of the drugs to be used in the study.
2. If Paracetamol contraindicated in severe hepatic impairment, or severe active hepatic disease.
3. If Diclofenac contraindicated in compromised renal function, increased risk of bleeding due to clotting disorder, an increased risk of bleeding, gastric ulcers, alcoholism.
4. If tramadol is contraindicated as in alcoholism, depression and drug abuse.
5. When a patient has a history of opioid abuse.
6. When a patient refuses to participate in the study.
7. When patient is unable to give consent.
8. Pregnancy.
9. If the patient has used conventional NSAIDs, Acetaminophen or Tramadol during the 6 hours before surgery,

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 176 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Pain score in post op period at 1 hour. | [1 hour]
  Pain score assessment at one hour by utilizing the Numeric Pain Intensity Scale (NPIS), score will be between 0-10.
Pain score in post op period at 6 hour. | [6 hour]
  Pain score assessment at six hour by utilizing the Numeric Pain Intensity Scale (NPIS), score will be between 0-10.
Pain score in post op period at 12 hour. | [12 hour]
  Pain score assessment at twelve hour by utilizing the Numeric Pain Intensity Scale (NPIS), score will be between 0-10.
Pain score in post op period at 24 hour. | [24 hour]
  Pain score assessment at twenty four hour by utilizing the Numeric Pain Intensity Scale (NPIS), score will be between 0-10.
Pain score in post op period at 48 hour. | [48 hour]
  Pain score assessment at forty eight hour by utilizing the Numeric Pain Intensity Scale (NPIS), score will be between 0-10.
Pain score in post op period at 72 hour. | [72 hour]
  Pain score assessment at seventy two hour by utilizing the Numeric Pain Intensity Scale (NPIS), score will be between 0-10.

SECONDARY OUTCOMES:
Patient Satisfaction | First 30 post-operative days
  Score on standardized evaluation of patient satisfaction at 7-days post-op. This was on a scale from 1) very dissatisfied to 5) very satisfied. Higher scores are better
4. Emergency visit for pain symptoms by the patients in the postoperative period after the discharge | First 30 post-operative days
  Number of times patients visited health facility for pain exacerbation
Hospital pain killers refill visits of patients for each category of analgesic used | 30 post-operative days
  Number of times patients visited health facility for refill pain killers medication

CONTACTS AND LOCATIONS:
Overall Officials: Nadeem Iqbal, FCPS*, Principal Investigator — Pakistan Kidney and Liver Institute
Locations (1):
- Pakistan Kidney and Liver Institute, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kang C, Shu X, Herrell SD, Miller NL, Hsi RS. Opiate Exposure and Predictors of Increased Opiate Use After Ureteroscopy. J Endourol. 2019 Jun;33(6):480-485. doi: 10.1089/end.2018.0796. Epub 2019 Feb 8. PMID 30618280
- [Background] Salaudeen GO, Afuwape OO, Eyelade OR, Olapade-Olaopa EO. Effectiveness of postoperative analgesia in the management of acute pain in day-case surgeries. Ann Afr Med. 2018 Jul-Sep;17(3):140-144. doi: 10.4103/aam.aam_53_17. PMID 30185683
- [Background] Klueh MP, Hu HM, Howard RA, Vu JV, Harbaugh CM, Lagisetty PA, Brummett CM, Englesbe MJ, Waljee JF, Lee JS. Transitions of Care for Postoperative Opioid Prescribing in Previously Opioid-Naive Patients in the USA: a Retrospective Review. J Gen Intern Med. 2018 Oct;33(10):1685-1691. doi: 10.1007/s11606-018-4463-1. Epub 2018 Jun 11. PMID 29948809
- [Background] Kasman AM, Schmidt B, Spradling K, Chow C, Hunt R, Wu M, Sockol A, Liao J, Leppert JT, Shah J, Conti SL. Postoperative opioid-free ureteroscopy discharge: A quality initiative pilot protocol. Curr Urol. 2021 Sep;15(3):176-180. doi: 10.1097/CU9.0000000000000025. Epub 2021 May 26. PMID 34552459
- [Background] Tam CA, Dauw CA, Ghani KR, Gunaseelan V, Kim T, Leavitt DA, Raisky J, Yan PL, Hollingsworth JM. New Persistent Opioid Use After Outpatient Ureteroscopy for Upper Tract Stone Treatment. Urology. 2019 Dec;134:103-108. doi: 10.1016/j.urology.2019.08.042. Epub 2019 Sep 16. PMID 31536742